CLINICAL TRIAL: NCT03058250
Title: Randomized Control Trial Comparing Routine Intraoperative Transesophageal Echocardiography During Radical Cystectomy to Standard of Care
Brief Title: Trial Comparing Routine Intraoperative Transesophageal Echocardiography During Radical Cystectomy to Standard of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB12-1694
Record Dates: First submitted 2017-02-13; First posted 2017-02-20 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Cardiac and Pulmonary Complications. Central Venous Line Insertion. Gastrointestinal Recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care, no intervention
- Transesophageal echocardiography (Active Comparator): Patients will have intraoperative transesophageal echocardiography along with standard of care for management.
  Interventions: Other: Transesophageal echocardiography

INTERVENTIONS:
Other: Transesophageal echocardiography
  Arms: Transesophageal echocardiography

SUMMARY:
This is a prospective randomized controlled trial looking at the utility of intraoperative transesophageal echocardiography (TEE) on clinical outcomes after radical cystectomy. Patients in the control group will have standard of care, patients in the TEE group will have standard of care and TEE monitoring throughout. Intraoperative and postoperative variables, such time to extubation, postoperative cardiac and pulmonary complications, intraoperative fluid and vasopressor use will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients have elective radical cystectomy at The University of Chicago Hospital.

Exclusion Criteria:

* Patient refusal, emergent surgery, preoperative mechanical ventilation, preoperative hemodynamic instability (intravenous vasopressor support), and/or esophageal/gastric pathology contraindicating insertion of the transesophageal echocardiography probe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative central venous line insertion | 1 day after study enrollment
postoperative return of bowel function via flatus or passage of stool | 5 days after study enrollment

SECONDARY OUTCOMES:
Decreased postoperative pulmonary and cardiac complications | approximately 5-7 days

IPD SHARING:
Plan to Share IPD: No